CLINICAL TRIAL: NCT00402883
Title: A Phase II Study of Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab in Patients With Unresectable Stage III Non-Small-Cell Lung Cancer
Brief Title: Chemotherapy, Radiotherapy and Bevacizumab in Patients With Unresectable Stage III Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to bevacizumab and chemoradiotherapy toxicity
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 134
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab; Pemetrexed; Radiotherapy; Folic Acid; Vitamin B 12; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Induction treatment included: carboplatin AUC=5, pemetrexed 500 mg/m2, and bevacizumab 15 mg/kg each administered intravenously weeks 1 and 4. Radiation was administered concurrently at a dose of 1.8 Gy/d weeks 1 to 7 to a total of 61.2 Gy per institutional guidelines. Consolidative therapy, following an 8-week break from chemoradiotherapy, included carboplatin AUC=6, pemetrexed 500 mg/m2, and bevacizumab 15 mg/kg each administered intravenously on week 16, repeated weeks 19 and 22. Folic acid (350 to 1,000 ug or equivalent) supplementation was administered orally beginning 1 to 2 weeks before the first dose of pemetrexed and continued daily until the patient discontinued study therapy. Vitamin B12(1,000ug) was administered by intramuscular injection 1 to 2 weeks before the first dose of study therapy and repeated every 9 weeks until the patient discontinued therapy.
  Interventions: Drug: Bevacizumab; Drug: Pemetrexed; Procedure: Radiotherapy; Other: Folic Acid; Other: vitamin B12; Drug: carboplatin

INTERVENTIONS:
Drug: Bevacizumab — 15mg/kg week 1, 4, 16, 19, 22, 25, 28, 31, 34, 37, 40, 43, 46, and 49.
  Other Names: Avastin
Drug: Pemetrexed — 500mg/m2 week 1, 4, 16, 19 and 22.
  Other Names: Alimta
Procedure: Radiotherapy — 1.8 Gy single daily fractions(Monday-Friday), to total dose 61.2 Gy (7 weeks)
  Other Names: RT
Other: Folic Acid — 350 to 1,000 ug or equivalent supplementation administered orally beginning 1 to 2 weeks before the first dose of pemetrexed and continued daily until the patient discontinues study therapy.
Other: vitamin B12 — 1,000ug administered by intramuscular injection 1 to 2 weeks before the first dose of study therapy and repeated every 9 weeks until the patient discontinues therapy.
Drug: carboplatin — AUC=5 administered intravenously weeks 1 and 4.

SUMMARY:
The purpose of this study is to see if this combination of chemotherapy plus radiation therapy and immunotherapy (with bevacizumab) expands treatment options for patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
The patients on this study will receive treatment in 3 stages of therapy.

The first stage is Induction Therapy. This therapy is 7 weeks long. Patients will receive bevacizumab followed by pemetrexed followed by carboplatin all by vein once a week in weeks 1 and 4. During Induction patients will also receive radiation therapy daily, Monday through Friday, for 7 weeks (weeks 1-7). This is followed by 2 weeks of rest. During this rest period patients will have scans done to see how their disease has responded to treatment.

The next stage of treatment is Consolidation Therapy. This stage is 10 weeks long. Patients will receive bevacizumab followed by pemetrexed followed by carboplatin all by vein once a week in weeks 10, 13 and 16. This is followed by 3 weeks rest. During week 19 patients will have scans to see how their disease has responded to treatment.

The last stage of treatment is Maintenance Therapy. Patients will receive bevacizumab alone by vein every 3 weeks. Treatment will be given every three weeks for up to 9 treatments. (week 45)

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed non-small cell lung cancer stage IIIA and selected stage IIIB
* Measurable or evaluable disease
* Be up and about and able to care for self
* Adequate kidney, liver and bone marrow function
* No prior treatment for this disease
* Must be able to give written informed consent
* Must be able to take folic acid, vitamin B12 and dexamethasone as described in the protocol
* Age 18 years or older

Exclusion Criteria:

* Stage IV or IIIB patients with pleural or pericardial effusions
* Stage IIIB disease with contralateral mediastinal nodes greater than 4cm
* Squamous cell predominant tumors
* Pregnant or lactating women
* Patients with active infections
* History of another cancer within the last 5 years with the exception of skin cancer or cervical carcinoma in situ
* History of stroke, transient ischemic attacks, or acute MI within the past 6 months or any other serious cardiovascular disease
* Symptoms of peripheral vascular disease
* History of neurological disease
* Recent history of blood in the sputum or vomitus
* Non-healing wounds, ulcer or long bone fractures
* History of bleeding problems or coagulation problems
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 6 months
* History of uncontrolled hypertension
* Chronic use of non-steroidal anti-inflammatory medication not allowed on this study

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Gainsville Hematology Oncology Associates, Gainesville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Wellstar Cancer Research, Marietta, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Oncology Hematology Care, Cincinnati, Ohio
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Yardley DA, Raefsky E, Patton J, Peacock N, Farley C, Burris HA 3rd, Greco FA. Tracheoesophageal fistula formation in patients with lung cancer treated with chemoradiation and bevacizumab. J Clin Oncol. 2010 Jan 1;28(1):43-8. doi: 10.1200/JCO.2009.24.7353. Epub 2009 Nov 9. PMID 19901100

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab: Induction treatment included: carboplatin AUC=5, pemetrexed 500 mg/m2, and bevacizumab 15 mg/kg each administered intravenously weeks 1 and 4. Radiation was administered concurrently at a dose of 1.8 Gy/d weeks 1 to 7 to a total of 61.2 Gy per institutional guidelines.
  Consolidative therapy, following an 8-week break from chemoradiotherapy, included carboplatin AUC=6, pemetrexed 500 mg/m2, and bevacizumab 15 mg/kg each administered intravenously on week 16, repeated weeks 19 and 22. Folic acid (350 to 1,000 ug or equivalent) supplementation was administered orally beginning 1 to 2 weeks before the first dose of pemetrexed and continued daily until the patient discontinued study therapy. Vitamin B12(1,000ug) was administered by intramuscular injection 1 to 2 weeks before the first dose of study therapy and repeated every 9 weeks until the patient discontinued therapy.
Period: Induction Therapy
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Started | 5
Completed | 5
Not Completed | 0
Period: Consolidation Therapy
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Started | 5
Completed | 5
Not Completed | 0
Period: Maintenance Therapy
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Started | 5
Completed | 5 (All 5 patients received limited maintenance therapy due to early trial closure.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Time Frame: 18 months
Population: No patients were analyzed due to the fact that the study ended early because of the formation of tracheoesophageal fistulas.
Arm/Group | Intervention
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate
Description: The objective benefit is defined as substantial shrinkage in tumor volume per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and is assessed by MRI or CT. Objective response = complete response + partial response. Complete Response (CR) is defined as the Disappearance of all target lesions; Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the date of study entry until the date of death
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Pemetrexed/Carboplatin/Radiotherapy and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5)
Chest Pain (Cardiac disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Difficulty swallowing (Gastrointestinal disorders) | 1 (1)
Transesophageal fistula (Gastrointestinal disorders) | 2 (2)
Dislodged PEG tube (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Non-ST elevation acute myocardial infarction (Cardiac disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Diffuse infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5)
Abdominal cramps (Gastrointestinal disorders) | 1 (1)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 (2)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (31)
Anxiety (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood in R nostril in morning (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CO2 (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (8)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Dehydration (Gastrointestinal disorders) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Discomfort (lower back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 4 (42)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Edema (lower extremities) (Blood and lymphatic system disorders) | 1 (2)
Esophageal strictures (Gastrointestinal disorders) | 1 (3)
Esophagitis (Gastrointestinal disorders) | 5 (30)
Fatigue (General disorders) | 5 (58)
Fever (General disorders) | 2 (2)
Gout - R finger (Metabolism and nutrition disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Hematologic - ANC (Blood and lymphatic system disorders) | 5 (22)
Hematologic - Hemoglobin (Blood and lymphatic system disorders) | 5 (39)
Hematologic - Platelets (Blood and lymphatic system disorders) | 5 (36)
Hematologic - WBC (Blood and lymphatic system disorders) | 5 (39)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage - nose (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hemorrhoid (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal bleeding (Gastrointestinal disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoxemia (Blood and lymphatic system disorders) | 2 (3)
Infection - sinus (Infections and infestations) | 1 (1)
Infection (pneumonia) (Infections and infestations) | 1 (2)
Interstitial fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (20)
Neuropathy - sensory (Nervous system disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 1 (5)
Pain - esophagus (Gastrointestinal disorders) | 3 (14)
Pain - shoulder blades (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - chest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - mediastinal (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 4 (9)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash - acneiform (scalp, neck) (Skin and subcutaneous tissue disorders) | 2 (5)
Rash - macular (arm) (Skin and subcutaneous tissue disorders) | 2 (5)
Rash - Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - erythema (Skin and subcutaneous tissue disorders) | 2 (8)
Shingles (Infections and infestations) | 1 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
TE fistula (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (10)
Weight loss (General disorders) | 4 (34)
Wheezes (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.